CLINICAL TRIAL: NCT03615599
Title: Cancer Epidemiology in Seventh-day Adventists
Brief Title: Plant-based Diets and Risk of Cancer in the Adventist Health Study-2
Acronym: AHS-2
Status: Active, not recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); World Cancer Research Fund International (Other); Ardmore Institute of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 48134; U01CA152939 (NIH); R01CA094594 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-08-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cancer, Breast; Cancer, Colorectal; Cancer, Prostate
Keywords: Seventh-day Adventists; vegetarian; mortality; cancer; dietary pattern; soy consumption; dairy consumption; plant-based
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat samples from a sample of the cohort (~2500) are stored from which DNA material may be extracted when a study requires such data. Other stored bio-specimens from a sample of the cohort include adipose tissue, urine, blood, sputum, stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seventh-day Adventists: This is a prospective cohort study of 96,000 members of the Seventh-day Adventists Church in the United States and Canada age 30 and older at the time of enrollment who are proficient in English language.

SUMMARY:
The Adventist Health Study-2 is a long-term study, exploring the links between lifestyle, diet, and disease outcomes among Seventh-day Adventists. More than 96,000 church members from the U.S. and Canada are participating in the current study, AHS-2, conducted by researchers at the Loma Linda University School of Public Health.

DETAILED DESCRIPTION:
The Adventist Health Study-2 (AHS-2) is a large national cohort of 96,000 Seventh-day Adventists in the U.S. and Canada. The study is searching for associations between diet and risk of common and medium frequency cancers (breast, prostate, colorectal, lung, uterus, pancreas, melanoma of skin). This cohort is unusual in that about half are vegetarian, many eat soy at Asian levels, and many have very low or absent dairy intake while others eat normal amounts of dairy. Thus observations on these people, many of whom have contrasting dietary habits, may provide insights about diet and cancer, so supporting dietary changes that could be readily adopted by many.

ELIGIBILITY:
Inclusion Criteria:

* Member of a Seventh-day Adventist church >30 years of age Ability to read English Live in the US or Canada

Exclusion Criteria:

* Less than 30 years of age
* Church members who did not complete the baseline questionnaire.
* Incarcerated or institutionalized people
* Non-English speakers

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample includes Seventh-day Adventist church members living in the USA and Canada who are 30 years and older, and who are sufficiently fluent in English to complete the lengthy lifestyle questionnaire. The study population is about 65% female. Approximately 25% of the cohort are Black/African Americans . Other ethnic minorities (e.g. Asian, Hispanic) are at much lower percentages (3-4 %).
Sampling Method: Non-Probability Sample
Enrollment: 96000 (Actual)
Dates: Start 2002-02-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incident cases of breast cancer among subjects with documented dietary habits. | Linkage with state cancer registries occurs periodically for 9 years, with first linkage at year 04 of study enrolment.
  Incident cases of breast cancer as found by linkage with state cancer registries will allow calculation of hazard ratios comparing extreme quintiles of dietary intakes. The focus is on meats, soy, and dairy intakes.

SECONDARY OUTCOMES:
Incident cases of prostate cancer among subjects with documented dietary intakes. | Linkage with state cancer registries occurs periodically for 9 years, with first linkage at year 04 of study enrolment.
  Incident cases of prostate cancer as found by linkage with state cancer registries will allow calculation of hazard ratios comparing extreme quintiles of dietary intakes. The focus is on meats, soy, and dairy intakes.

OTHER OUTCOMES:
Incident cases of colorectal cancer among subjects with documented dietary habits. | Linkage with state cancer registries occurs periodically for 9 years, with first linkage at year 04 of study enrolment.
  Incident cases of colorectal cancer as found by linkage with state cancer registries will allow calculation of hazard ratios comparing extreme quintiles of dietary intakes. The focus is on meats, soy, and dairy intakes.

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Fraser, MD,PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers must write a proposal describing how the data will be used and submit it to the Adventist Health Study data sharing committee for approval.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: on-going
Access Criteria: Data access will be given upon approval of proposal by the AHS-2 Review Committee.
URL: http://www.ahs2.org

REFERENCES:
- [Background] Butler TL, Fraser GE, Beeson WL, Knutsen SF, Herring RP, Chan J, Sabate J, Montgomery S, Haddad E, Preston-Martin S, Bennett H, Jaceldo-Siegl K. Cohort profile: The Adventist Health Study-2 (AHS-2). Int J Epidemiol. 2008 Apr;37(2):260-5. doi: 10.1093/ije/dym165. Epub 2007 Aug 27. No abstract available. PMID 17726038
- [Derived] Fraser GE, Jacobsen BK, Knutsen SF, Mashchak A, Lloren JI. Tomato consumption and intake of lycopene as predictors of the incidence of prostate cancer: the Adventist Health Study-2. Cancer Causes Control. 2020 Apr;31(4):341-351. doi: 10.1007/s10552-020-01279-z. Epub 2020 Feb 25. PMID 32100191